CLINICAL TRIAL: NCT01247844
Title: Evaluation of Healing at Three Time Intervals and Potential for Spontaneous Detachment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: Kenya National AIDS & STI Control Programme (Other); Ministry of Medical Services, Kenya (Other); EngenderHealth (Other); Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 10214
Record Dates: First submitted 2010-09-07; First posted 2010-11-24 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Male Circumcision
Keywords: adult Males; circumcision; HIV prevention; device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Day 7 (Other): removal of Shang Ring at 7 days
  Interventions: Device: Shang Ring
- Day 14 (Other): removal of Shang Ring at 14 days
  Interventions: Device: Shang Ring
- Day 21 (Other): removal of Shang Ring at 21 days
  Interventions: Device: Shang Ring

INTERVENTIONS:
Device: Shang Ring — The Shang Ring is a sterile device consisting of two concentric medical grade plastic rings: an inner ring with a silicone band and an outer, hinged ring. The inner ring fits inside the outer ring which will lock when snapped together. The Shang Ring comes in multiple sizes. The appropriate size is determined through use of a measuring strip. The man must return to the clinic for device removal. To remove the device, the outer ring locking mechanism is broken open using a tool that is similar to a scalpel handle. Then, a pair of special scissors, specifically designed for this purpose, is used to remove the inner ring after healing

SUMMARY:
The objective of this research study is to evaluate the safety and acceptability of the Shang Ring method of medical male circumcision. The Shang Ring is a new circumcision device with a potential role in the safe and cost-effective delivery of circumcision services. The device, developed in China, consists of two concentric plastic rings. Following a ring penile block, the smaller ring is fitted at the base of the coronal sulcus. The foreskin is everted over the inner ring and the larger outer ring is secured over the inner ring. The foreskin is excised and several nicks are made on the incision line to prevent formation of a constricting, circumferential scab. No suturing is required.

In this study, the investigators will evaluate wound healing of men randomized to removal of the Shang Ring at one of three different points in time (Days 7, 14 or 21). Leaving the device on for 14 or 21 days constitutes extended wear of the device.

Sites: Homa Bay District Hospital, Nyanza Province, Kenya

DETAILED DESCRIPTION:
The objective of this research study is to evaluate the safety and acceptability of the Shang Ring method of medical male circumcision. The Shang Ring is a new circumcision device with a potential role in the safe and cost-effective delivery of circumcision services. The device, developed in China, consists of two concentric plastic rings. Following a ring penile block, the smaller ring is fitted at the base of the coronal sulcus. The foreskin is everted over the inner ring and the larger outer ring is secured over the inner ring. The foreskin is excised and several nicks are made on the incision line to prevent formation of a constricting, circumferential scab. No suturing is required.

In this study, we will evaluate wound healing of men randomized to removal of the Shang Ring at one of three different points in time (Days 7, 14 or 21). Leaving the device on for 14 or 21 days constitutes extended wear of the device.

Although male circumcision has a demonstrated protective effect against HIV transmission, currently available surgical techniques and devices have limitations for widespread deployment in resource-poor areas. High costs and scarcity of trained providers hinder access to male circumcision services in resource-poor areas. Its simple design sets the Shang Ring apart from other male circumcision techniques. The Shang Ring has the potential for safe, effective and inexpensive delivery of male circumcision by trained healthcare personnel in HIV endemic countries.

ELIGIBILITY:
Inclusion Criteria:

* Must be aged 18 and 54 years;
* Must be uncircumcised (on examination);
* Must be in good general health;
* Must be HIV sero-negative, with documentation of testing no mor than one week before the procedure;
* Must be free of genital ulcerations or other visible signs of sexually transmissible infections(STI) on examination;
* Must be able to understand study procedures and requirements of study participation;
* Must agree to return to the healthcare facility for the full schedule of follow-up visits after his circumcision;
* Must freely consent to participate in the study and sign a written informed consent form;
* Must have a cell phone or access to a cell phone; and,
* Must agree to provide the study staff with an address, phone number, or other locator information while participating in the research study.

Exclusion Criteria:

* Has a known allergy or sensitivity to lidocaine or other local anesthesia;
* Takes a medication that would be a contraindication for elective surgery, such as an anticoagulant or steroid;
* Has an active genital infection, anatomic abnormality or other condition, which in the opinion of the surgeon, prevents the man from undergoing a circumcision;
* Has known bleeding/clotting disorder (e.g. hemophilia); and,
* Has thalassemia (an inherited autosomal recessive blood disease).

Ages: 18 Years to 54 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Asses healing time | six weeks
  Assess healing time from date of circumcision
spontaneous detachment of device | 21 days
  Spontaneous detachment from date of circumcision to three weeks post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Marc Goldstein, M.D., Study Chair — Weill Cornell Medical College, NY, USA; Mark Barone, DVM; MS, Study Chair — EngenderHealth, NY, USA; Philip S. Li, MD, Principal Investigator — Weill Medical College of Cornell University; Puneet Masson, MD, Principal Investigator — Weill Medical College of Cornell University; Paul Perchal, MA, Principal Investigator — EngenderHealth; Jared Moguche, MB ChB, Principal Investigator — EngenderHealth; Quentin Awori, MB ChB, Principal Investigator — Engender Health; Peter Cherutich, MB ChB MPH, Principal Investigator — National AIDS/STD Control Programme, Nairobi, Kenya; Nicholas Muraguri, MB ChB MPH, Principal Investigator — National AIDS/STD Control Programme; John Masasabi Wekesa, MB ChB MMed, Principal Investigator — Ministry of Medical Services Nairobi Kenya; Robert Otieno Simba, MMed, Principal Investigator — Homa Bay District Hospital
Locations (1):
- Homa Bay District Hospital, Homa Bay, Nyanza, Kenya